CLINICAL TRIAL: NCT00984386
Title: A Single Site, Placebo and Standard Care Controlled, Double Blind, Randomised Trial to Investigate the Efficacy of Four Doses of Zesteem in Accelerating Early Wound Healing of Punch Biopsy Skin Wounds.
Brief Title: Investigation of the Efficacy of Zesteem in Accelerating Early Wound Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1002-028
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound-healing
Keywords: Cicatrix; Scar; Wound-healing; Zesteem; 17β-Estradiol; RN1002
MeSH Terms: conditions — Cicatrix | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal Zesteem (Experimental)
  Interventions: Drug: Zesteem
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zesteem — Intradermal Zesteem, 0.02μg/100μl administered once before punch biopsy
  Other Names: 17β-Estradiol; RN1002
  Arms: Intradermal Zesteem
Drug: Zesteem — Intradermal Zesteem, 0.1μg/100μl administered once before punch biopsy
  Other Names: 17β-Estradiol; RN1002
  Arms: Intradermal Zesteem
Drug: Zesteem — Intradermal Zesteem, 0.2μg/100μl administered once before punch biopsy
  Other Names: 17β-Estradiol; RN1002
  Arms: Intradermal Zesteem
Drug: Zesteem — Intradermal Zesteem, 0.4μg/100μl administered once before punch biopsy
  Other Names: 17β-Estradiol; RN1002
  Arms: Intradermal Zesteem
Drug: Placebo — Intradermal placebo, 100μl administered once before punch biopsy
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate early wound healing of one application of four different doses of intradermal Zesteem (17β-Estradiol) in male subjects and female subjects two years post-menopausal.

DETAILED DESCRIPTION:
Each subject received a total of six, 3mm punch biopsy wounds; three wounds to the upper inner aspect of each arm. Each punch biopsy site was randomly allocated to receive one of six treatments: Zesteem (0.02μg, 0.1μg, 0.2μg and 0.4μg/100μl), Placebo (vehicle), and Standard Care (moist wound healing dressings) only.

Zesteem and Placebo were administered to marked, anaesthetised sites, by intradermal injection 10 to 30 minutes before wounding. Sites randomised to receive Standard Care only received no additional treatment before wounding. After wounding, all sites received moist wound healing dressings (Standard Care).

Three days after wounding, all biopsy sites were anaesthetised and the wounds excised using a 5mm punch biopsy, for histological analysis. The Investigator closed all excision sites using sutures and Steri-strips to achieve a cosmetically acceptable result. Subjects attended a post-trial follow-up visit (13-18 days after dosing) where their sutures were removed and final safety assessments were performed.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-85 years, and female subjects who are at least two years postmenopausal (quantified by a serum test result of estradiol <90 pmol/L and FSH > 31 IU/L) who have given written informed consent
* Subjects with a BMI within the permitted range for their height using Quetelet's index-weight (kg)/height² (m). The permitted index is 15-55 kg/m2
* Subjects with, in the opinion of the investigator, clinically acceptable results for laboratory safety tests performed within 28 days of the first trial dose administration

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have history or evidence of hypertrophic or keloid scarring
* Subjects with tattoos or previous scars within 3cm of the area to be biopsied
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring
* Subjects who have had surgery in the area to be biopsied within one year of the first dosing day
* Subjects with a history of a bleeding disorder
* Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial
* Subjects with any clinically significant medical condition or history that would impair wound healing including: significant rheumatoid arthritis, chronic renal impairment significant for their age, significant hepatic impairment (LFTs >3 times upper limit of normal), congestive heart failure, current active malignancy or history of malignancy in the last 5 years, immunosuppression or chemotherapy within the last 12 months, a history of radiotherapy or diabetes mellitus
* Subjects with a history of hypersensitivity to any of the drugs or dressings used in this trial
* Subjects who are taking, or have taken any investigational product or participated in a clinical trial in the three months prior to first trial dose administration
* Subjects who are taking regular, continuous, oral corticosteroid therapy
* Subjects undergoing investigations or changes in management for an existing medical condition
* Subjects with a history of drug abuse
* Subjects with a positive drugs of abuse test for cocaine, amphetamines, methamphetamines, opiates or benzodiazepines during the screening period
* Subjects who, in the opinion of the investigator, are unlikely to complete the trial for whatever reason
* Female subjects who are currently taking any form of hormone replacement therapy or contraceptive medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To assess acceleration of early wound healing in male and postmenopausal female subjects following administration of intradermal Zesteem. The primary trial endpoint will be the distance travelled by the epithelium over the biopsy site. | Day 3

SECONDARY OUTCOMES:
To assess safety and tolerability of intradermal Zesteem in male and post-menopausal female subjects. | 13-18 Days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duncan, Principal Investigator — Renovo
Locations (1):
- Renovo Clinical Trials Unit, Manchester, United Kingdom